CLINICAL TRIAL: NCT02612857
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial of IMO-8400 in Patients With Dermatomyositis
Brief Title: Trial of IMO-8400 in Adult Patients With Dermatomyositis
Acronym: 8400-211
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8400-211
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Dermatomyositis
Keywords: dermatomyositis; IMO-8400; Pioneer
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): normal saline subcutaneous injections once a week for 24 weeks.
  Interventions: Drug: Placebo
- IMO-8400 Dose Group 1 (Experimental): IMO-8400 Dose Group 1 subcutaneous injections once a week for 24 weeks.
  Interventions: Drug: IMO-8400 Dose Group 1
- IMO-8400 Dose Group 2 (Experimental): IMO-8400 Dose Group 2 subcutaneous injections once a week for 24 weeks.
  Interventions: Drug: IMO-8400 Dose Group 2

INTERVENTIONS:
Drug: IMO-8400 Dose Group 1 — IMO-8400 Dose 1 subcutaneous injections once a week for 24 weeks.
  Arms: IMO-8400 Dose Group 1
Drug: IMO-8400 Dose Group 2 — IMO-8400 Dose 2 subcutaneous injections once a week for 24 weeks.
  Arms: IMO-8400 Dose Group 2
Drug: Placebo — normal saline subcutaneous injections once a week for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine how safe and effective IMO-8400 is in adults with dermatomyositis.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of IMO-8400 in adults with active dermatomyositis (DM).

ELIGIBILITY:
Inclusion Criteria:

* Has definite or probable DM based on the criteria of Bohan and Peter
* Has a Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)-Activity score ≥15
* Patients with muscle weakness are eligible; however having muscle weakness is not mandatory.
* Study participants must have a diagnostic evaluation for cancer if the diagnosis of DM was within 2 years prior to the Screening Visit

Exclusion Criteria:

* Has ongoing severe dysphagia (e.g., requires a feeding tube) for the 3 months prior to Screening
* Has known hypersensitivity to any oligodeoxynucleotide
* Has a history of drug or alcohol abuse within one year of screening, or evidence of drug abuse by urine drug screening
* Has body weight >140 kg
* Has a diagnosis of Juvenile DM, IBM, drug-induced toxic myopathy, metabolic myopathy, dystrophy, cancer-associated DM, or connective tissue disease-associated DM (e.g., overlap syndrome)
* Has received one or more of following prohibited treatments within the interval noted prior to Screening (Visit 1):

  1. Rituximab within 24 weeks (Note: patients who received rituximab are only eligible for inclusion if B-cell counts are confirmed to be within normal limits)
  2. Intravenous corticosteroids within 12 weeks
  3. Antimalarials (e.g., hydroxychloroquine) within 36 weeks
  4. Topical corticosteroids (excluding scalp) within 2 weeks
* Has evidence of or has required treatment for cancer (except for treated, non-invasive carcinoma of the skin or cured cervical carcinoma-in-situ) within 5 years
* Has interstitial lung disease requiring the use of supplemental oxygen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Horobin, MD, Study Director — Idera Pharmaceuticals
Locations (20):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - Stanford Hospital and Clinics, Stanford, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Northwell Health, Great Neck, New York
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Vermont College of Medicine, Burlington, Vermont
- University of Debrecen, Debrecen, Hungary
- United Kingdom (2):
  - MRC/ARUK Institute of Ageing and Chronic Disease, University of Liverpool, Liverpool
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IMO-8400 Dose Group 1: IMO-8400 Dose Group 1 subcutaneous injections once a week for 24 weeks.
  IMO-8400 Dose Group 1: 0.6mg/kg IMO-8400 Dose 1 subcutaneous injections once a week for 24 weeks.
- IMO-8400 Dose Group 2: IMO-8400 Dose Group 2 subcutaneous injections once a week for 24 weeks.
  IMO-8400 Dose Group 2: 1.8mg/kg IMO-8400 Dose 2 subcutaneous injections once a week for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | IMO-8400 Dose Group 1 | IMO-8400 Dose Group 2
Started | 11 | 9 | 10
Completed | 8 | 5 | 6
Not Completed | 3 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IMO-8400 Dose Group 1 | IMO-8400 Dose Group 2 | Total
Number analyzed (Participants) | 11 | 9 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (10.55) | 48.3 (14.23) | 54.6 (14.12) | 51.5 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 9 | 23
  Male | 4 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 10 | 8 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 2 | 1 | 2 | 5
  United States | 8 | 8 | 8 | 24
  United Kingdom | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Safety and Tolerability of IMO-8400 in Adult Subjects With DM
Description: Number of participants with different types of Treatment Emergent Adverse Events
Time Frame: 28 weeks (24 weeks treatment + 4 weeks follow up)
Measure: Number; unit: participants
Arm/Group | Placebo | IMO-8400 Dose Group 1 | IMO-8400 Dose Group 2
Number analyzed (Participants) | 11 | 9 | 10
participants
  TEAE Severity Mild | 6 | 4 | 2
  TEAE Severity Moderate | 4 | 3 | 6
  TEAE Severity Severe | 1 | 2 | 2
  TEAE Causality Probably Related | 3 | 9 | 9
  TEAE Causality Possibly Related | 3 | 0 | 1
  TEAE Causality Not Related | 5 | 0 | 0
  Injection Site Reaction AE | 2 | 8 | 10
  Serious TEAE | 0 | 0 | 1
  TEAE Leading to Treatment Discontinuation | 1 | 3 | 1
  TEAE Leading to Death | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in CDASI (Cutaneous Disease and Activity Severity Index) Activity Score
Description: Change from baseline in mCDASI (Cutaneous Disease and Activity Severity Index) v2-Activity score as measured at Visits 2, 6, 10, 14, 18, 22 and 26 (EOT/ Week 25). Index is Clinician administered one page instrument designed to evaluate the cutaneous manifestations of DM. CDASI yields a total score that captures overall disease state, an activity score (range:0-100) that reflects the current inflammatory state of disease and a damage score (range: 0-32). The CDASI includes separate measurements for disease activity and damage and yields a total score that captures overall disease state, an activity score that reflects the current inflammatory state of disease, and a damage score. Decreases in CDASI scores are indicative of improvement. In this study, Activity Scores were measured. The scores below are averaged.
Time Frame: 28 weeks (24 weeks treatment + 4 weeks follow up)
Population: Some patients did not complete all visits
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | IMO-8400 Dose Group 1 | IMO-8400 Dose Group 2
Number analyzed (Participants) | 11 | 9 | 10
units on a scale
  Baseline | 30.1 [29.60 to 30.56] | 31.3 [30.72 to 31.79] | 30.7 [30.20 to 31.22]
  Visit 6: number analyzed (Participants) | 11 | 8 | 10
  Visit 6 | 28.0 [25.23 to 30.76] | 28.5 [25.27 to 31.66] | 27.8 [24.91 to 30.71]
  Visit 10: number analyzed (Participants) | 10 | 7 | 9
  Visit 10 | 27.7 [23.66 to 31.83] | 30.4 [25.54 to 35.26] | 25.7 [21.40 to 30.07]
  Visit 14: number analyzed (Participants) | 10 | 7 | 7
  Visit 14 | 28.9 [24.46 to 33.35] | 29.4 [24.17 to 34.70] | 21.6 [16.75 to 26.51]
  Visit 18: number analyzed (Participants) | 10 | 5 | 8
  Visit 18 | 30.5 [25.71 to 35.22] | 26.0 [19.98 to 32.09] | 22.4 [17.24 to 27.63]
  Visit 22: number analyzed (Participants) | 7 | 6 | 8
  Visit 22 | 26.6 [20.59 to 32.61] | 25.3 [18.40 to 32.13] | 24.6 [18.39 to 30.82]
  Visit 26: number analyzed (Participants) | 8 | 6 | 6
  Visit 26 | 26.0 [20.97 to 31.04] | 22.1 [16.19 to 28.01] | 23.0 [17.38 to 28.61]
  Across Visit | 28.3 [24.74 to 31.77] | 27.6 [23.41 to 31.72] | 25.1 [21.36 to 28.90]

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Placebo | IMO-8400 Dose Group 1 | IMO-8400 Dose Group 2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 11/11 | 9/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | IMO-8400 Dose Group 1 (N=9) | IMO-8400 Dose Group 2 (N=10)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | IMO-8400 Dose Group 1 (N=9) | IMO-8400 Dose Group 2 (N=10)
Injection Site Erythema (General disorders) | 1 | 7 | 10
Injection Site Pain (General disorders) | 0 | 6 | 7
Injection Site Induration (General disorders) | 0 | 5 | 5
Injection Site Pruritis (General disorders) | 0 | 3 | 5
Injection Site Bruising (General disorders) | 0 | 2 | 4
Fatigue (General disorders) | 0 | 3 | 2
Injection Site Vesicles (General disorders) | 0 | 0 | 3
Injection Site Haematoma (General disorders) | 1 | 1 | 0
Injection Site Rash (General disorders) | 0 | 0 | 2
Malaise (Gastrointestinal disorders) | 0 | 1 | 1
Application Site Alopecia (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 0
Feeling Hot (General disorders) | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1 | 0
Injection Site Discolouration (General disorders) | 0 | 1 | 0
Injection Site Exfoliation (General disorders) | 0 | 0 | 1
Injection Site Haemorrhage (General disorders) | 0 | 1 | 0
Injection Site Swelling (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Dermatomyositis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Distention (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Faeces Soft (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0
Genital Herpes Simplex (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Antisynthetase syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Burning Sensation (Nervous system disorders) | 0 | 0 | 1
Head Discomfort (Nervous system disorders) | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Complement factor C3 decreased (Investigations) | 0 | 2 | 1
Anti-platelet antibody positive (Investigations) | 0 | 2 | 0
Weight Increased (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Double stranded DNA antibody positive (Investigations) | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat Lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Psychosomatic Disease (Psychiatric disorders) | 0 | 0 | 1
Hot Flush (Vascular disorders) | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Benign Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT02612857/SAP_000.pdf
  • Study Protocol (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT02612857/Prot_001.pdf